CLINICAL TRIAL: NCT06915207
Title: Integrative Medical Care For Adult Depression: A One Year Pilot Project
Brief Title: Adult Depression and Integrative Medical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Anne Leis, Principal Investigator, University of Saskatchewan
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USaskatchewan-CH&E
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Depression
Keywords: adults; Depression; Integrative medical care; quasi-experimental design
MeSH Terms: conditions — Depression | interventions — Counseling; Nutritional Status

STUDY DESIGN:
Intervention Model Description: Longitudinal over 1 year
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care for depression (No Intervention): Medication for depression
- Intervention (Active Comparator): Integrative medical care
  Interventions: Dietary Supplement: Counselling, behavioural, nutrition

INTERVENTIONS:
Dietary Supplement: Counselling, behavioural, nutrition — integrative medical care delivered by one physician and referral to other health professionals as appropriate
  Arms: Intervention

SUMMARY:
The goal of this quasi-experimental study is to learn if integrative medical care works to treat depression in adults and compare it to usual medical care. The main question it aims to answer is to find out whether integrative medical care is equal or better to usual medical care in treating depressed adults over one year.

Participants attended five data collection visits which occurred at baseline, 3, 6, 9 and 12 months. At each visit, they completed questionnaires and had a small blood sample drawn. They were also asked to keep a diary of their symptoms and what they did between visits. They brought a calendar summary with a saliva sample at visits 2 to 5.

ELIGIBILITY:
Inclusion Criteria:

* experiencing depressive symptoms as defined by a Centre for Epidemiologic Studies-Depression (CES-D) scale score of 16 or higher as categorized by Lewinsohn et al.
* willing to commit to five study visits over one year.

Exclusion Criteria:

* substance abuse
* pregnancy
* non-depression neurological problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in depression | one year
  as measured by the Beck Depression Inventory (BDI) test. It has a continuous range of whole number scores from 0-63 that correspond to four categories of depression: minimal (0-13), mild (14-19), moderate (20-28) and severe (29-63)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Leis, PhD, Principal Investigator — University of Saskatchewan; Shirley Maltman, MD, Study Chair — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
This is a small pilot study
Supporting Information: CSR
Time Frame: within 3 months